CLINICAL TRIAL: NCT02457533
Title: Active Support to Patient With COLD
Brief Title: Case Management - Active Telephone Support to Patients With COLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Sjælland (Other)
Collaborators: Health Navigator, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CM1
Record Dates: First submitted 2015-04-23; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: COLD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Only SF-36 and CAT
- Active (Active Comparator): Lifestyle behavioral. Health plan, telephone support
  Interventions: Behavioral: Lifestyle behavioral. Health plan, telephone support

INTERVENTIONS:
Behavioral: Lifestyle behavioral. Health plan, telephone support — 'Lifestyle behavioral. Health plan, telephone support'
  Arms: Active

SUMMARY:
To investigate the effects of patient counseling by telephone on Quality of Life and the use of Health care system.

DETAILED DESCRIPTION:
By analyzing patient data, patients with risk of high consumption of the Health system are identified.

These patients are invited to take part in the study. If the patient accept the invitation, oral and written information of the study is given. If the patient give informed consent to participate, the inclusion and exclusion criteria and the patient record are examined.

If the patient meet the criteria the patient is randomized to active treatment or control 1:1.

Patient in the Intervention Group have a in depth interview of Health and social status and possible interventions are planned. Following that, the patient is contacted by telephone on weekly intervals for 6 to 9 months.

Patients in both Groups fill out questionaire Short-Form Health Survey-36 (SF-36) and COPD Assessment Test (COPD) and the consumption of Health care is monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patient living in The Zealand Region.
* A COLD-related contact with hospital with-in 6 months.
* Predicted to be in high risk of new hospital admission.

Exclusion Criteria:

* Dementia.
* Psychosis.
* Drug-addiction.
* Cancer with metastasis.
* Terminal illness.
* Language difficulties demanding translator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-10 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Life questionnaire SF-36 (Short-Form Health Survey) | Participants will be followed an expected avarage of 6 months

SECONDARY OUTCOMES:
Analysis of patients use of Health Care system | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Knud Rasmussen, MD DMSci, Principal Investigator — Region of Zealand
Locations (1):
- Regional Research, Roskilde, Denmark